CLINICAL TRIAL: NCT06930092
Title: RestoratIon of Myocardial Function by PeRcutaneous cOronary interVEntion in Patients With Ischemic CardioMyoPathy
Acronym: IMPROVE-ICMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Seoul National University Boramae Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2411-106-1590; Not yet assigned (Other Grant/Funding Number: Chong Kun Dang); Not yet assigned (Other Grant/Funding Number: Dotter)
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Ischemic Cardiomyopathy
Keywords: percutaneous coronary intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physiology-and imaging-guided PCI (Experimental): The goal is to achieve functional complete revascularization of major coronary arteries and their branches with diameters ≥2.5 mm. For lesions with ≥50% diameter stenosis, fractional flow reserve (FFR) measurement is mandatory. However, for severely stenotic lesions (>90%), revascularization may proceed at the operator's discretion without FFR assessment. In addition, intravascular ultrasound (IVUS) should be utilized during revascularization procedures and serve as an additional criterion for decision-making.
  All patients in the intervention group will receive optimal medical therapy identical to that provided to the optimal medical therapy group following PCI.
  Interventions: Procedure: Physiology-and imaging-guided PCI
- Optimal medical treatment (Active Comparator): All study participants will receive guideline-directed medical therapy, including an angiotensin receptor-neprilysin inhibitor (ARNi) or an angiotensin-converting enzyme inhibitor (ACEi) or angiotensin receptor blocker (ARB), a beta-blocker (carvedilol or bisoprolol), an aldosterone antagonist, and an SGLT2 inhibitor (empagliflozin or dapagliflozin). Medications will be administered even at low doses, as tolerated based on the patient's clinical status. Antiplatelet agents and statins will be maintained throughout the study period, and ezetimibe or PCSK9 inhibitors may be added as needed.
  In addition, appropriate treatment will be provided for major cardiovascular risk factors such as hypertension, diabetes, and hyperlipidemia. Coexisting arrhythmias will be managed according to their respective guidelines. In the case of atrial fibrillation, active rate and rhythm control strategies will be implemented.
  Interventions: Drug: Optimal medical treatment

INTERVENTIONS:
Procedure: Physiology-and imaging-guided PCI — The criteria for performing revascularization are as follows
  1. Lesions with ≥50% diameter stenosis and FFR ≤ 0.80, or lesions with severe stenosis (>90%)
  2. In vessels meeting the above criteria, IVUS findings consistent with either:
     * Minimum lumen area (MLA) ≤ 3 mm²
     * 3 mm² < MLA ≤ 4 mm² and plaque burden >70%
  For all target vessels and lesions identified for intervention, optimal revascularization should be pursued. The criteria for optimal revascularization are as follows, and operators are encouraged to achieve them:
  1. Post-PCI FFR > 0.86 in all treated vessels is recommended, with a minimum threshold of post-PCI FFR > 0.80 to achieve functional complete revascularization.
  2. Post-PCI ΔFFR (defined as [FFR at stent distal edge] - [FFR at stent proximal edge]) < 0.05 is recommended.
  3. On IVUS, achieving a minimum stent area (MSA) > 5.5 mm² and MSA/average reference lumen > 80% is recommended.
  Arms: Physiology-and imaging-guided PCI
Drug: Optimal medical treatment — All study participants will receive guideline-directed medical therapy. Even for patients assigned to the optimal medical therapy group, revascularization may be performed during follow-up if clinically indicated. If such a decision is made prior to the primary endpoint assessment, a gadolinium-enhanced cardiac MRI will be performed at the time of consideration to reassess myocardial viability.
  Arms: Optimal medical treatment

SUMMARY:
To compare the effects of physiology- and imaging-guided PCI combined with optimal medical therapy (OMT) versus OMT alone on the recovery of left ventricular systolic function in patients with ischemic cardiomyopathy and multivessel coronary artery disease.

DETAILED DESCRIPTION:
This study is a prospective, open-label, randomized, multicenter trial to test the safety and efficacy of physiology- and imaging-guided complete revascularization with PCI combined with optimal medical therapy (OMT) versus OMT alone on the recovery of left ventricle ejection fraction (LVEF) in patients with ischemic cardiomyopathy and multivessel coronary artery disease.

The primary hypothesis is that physiology- and imaging-guided complete revascularization with PCI combined with OMT will show greater improvements in LV systolic function at 6 months after randomization compared with OMT alone.

Patients with left ventricular ejection fraction (LVEF) less than 40% on echocardiography will undergo gadolinium-enhanced cardiac MRI to determine the underlying cause of cardiac dysfunction and assess the presence of viable myocardium. Among patients suspected of having ischemic cardiomyopathy, those who provide informed consent will be considered for enrollment. Eligible patients undergoing invasive coronary angiography and meeting inclusion and exclusion criteria will be randomly assigned to either: a group receiving physiology- and imaging-guided PCI in combination with optimal medical therapy, or a group receiving optimal medical therapy alone.

Improvement in LVEF will be evaluated using follow-up gadolinium-enhanced cardiac MRI at 6 months. Clinical outcomes will be assessed at 6 and 12 months, and long-term outcomes will be analyzed through 36-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 19 years
* Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving invasive physiologic or imaging evaluation and PCI and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
* Subject with LV ejection fraction <40% from cardiac MRI
* Subject with multivessel disease in major epicardial coronary artery disease or their major branches (vessel size of 2.5 mm or more than 2.5mm) considering coronary revascularization

Exclusion Criteria:

* Subjects with more than 50% transmural extent of infarction on GE-MRI in more than 25% of the dysfunctional myocardial segments
* Subject with suspicious of other cardiomyopathy (dilated cardiomyopathy, hypertrophic cardiomyopathy etc.)
* Subject with recent myocardial infarction within 4 weeks
* Subject with recent fatal arrhythmia (VT or VF) within 4 weeks
* Subject with hemodynamically unstable state
* Subject with complex coronary artery lesions, such as chronic total occlusions, in which complete revascularization is considered unfeasible
* Subject for whom coronary artery bypass surgery is prioritized over coronary artery intervention
* Subject with severe valvular heart disease requiring open heart surgery
* Subject with history of coronary artery bypass surgery or valve surgery
* Subject with expected life expectancy of less than 1 year
* Subject considered ineligible for this study based on the investigator's discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
LV ejection fraction from GE-MRI | At 6 months after randomization
  LV ejection fraction from gadolinium-enhanced MRI

SECONDARY OUTCOMES:
Changes in the transmural extent of myocardial infarction from GE-MRI | At 6 months after randomization
  Changes in the transmural extent of myocardial infarction from GE-MRI
Number of improved dysfunctional myocardial segments from GE-MRI | At 6 months after randomization
  Number of improved dysfunctional myocardial segments from GE-MRI
Changes in the LV chamber size from GE MRI | At 6 months after randomization
  Changes in the LV chamber size from GE MRI
LV ejection fraction from echocardiography | At 6 months and 12 months after randomization
  LV ejection fraction from echocardiography
Number of improved dysfunctional myocardial segments from echocardiography | At 6 months and 12 months after randomization
  Number of improved dysfunctional myocardial segments from echocardiography
Changes in the LV chamber size change from echocardiography | At 6 months and 12 months after randomization
  Changes in the LV chamber size change from echocardiography
All-cause death | At 6 months, 12 months, and 36 months after randomization
  death from any cause
Cardiovascular death | At 6 months, 12 months, and 36 months after randomization
  death from cardiovascular cause
Non-fatal myocardial infarction | At 6 months, 12 months, and 36 months after randomization
  Non-fatal myocardial infarction
Unplanned revascularization | At 6 months, 12 months, and 36 months after randomization
  Unplanned revascularization
Hospitalization for heart failure | At 6 months, 12 months, and 36 months after randomization
  Hospitalization for heart failure
EuroQol 5-Dimension 5-Level Questionnaire | At 6 months, 12 months, and 36 months after randomization
  EuroQol 5-Dimension 5-Level Questionnaire
Brain natriuretic peptide (BNP or NT-Pro BNP) level | At 6 months, 12 months, and 36 months after randomization
  Brain natriuretic peptide (BNP or NT-Pro BNP) level

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Chongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: Yes
The deidentified data will be shared after publication of first manuscript
Time Frame: Data will be available within 12 months of study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement